CLINICAL TRIAL: NCT04526847
Title: Effectiveness of Intermittent Fasting Compared to Continuous Energy Restriction on Body Weight Loss Among Overweight/Obese Adults: a Randomized Controlled Trial
Brief Title: Intermittent Fasting Compared to Continuous Energy Restriction on Body Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Armed Police Force Hospital, Nepal (Other Government)
Responsible Party: Principal Investigator, Dev Ram Sunuwar, Principal Investigator, Armed Police Force Hospital, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Intermittent Fasting
Record Dates: First submitted 2020-08-19; First posted 2020-08-26 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Overweight and Obesity
Keywords: Intermittent fasting; energy restriction; weight loss; cardiometabolic risk markers; Nepal
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting; Weight Loss | interventions — Population Groups; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: The proposed study is a parallel arm, randomized controlled trial compare two different dietary patterns: 1) intermittent energy-restriction (IER) diet also known as intermittent fasting (5:2 eating pattern: 5 days of habitual intake and 2 very low energy diet on two non-consecutive days (Mondays and Thursdays) per week, and 2) Continuous (daily) energy-restricted diet (CER) on the reduction of body weight, and cardiometabolic risk factors among overweight/obese Nepalese population (Figure 2). This study will adopt a parallel randomized trial design with an equal allocation of participants between the IER and CER arm. The participants will be recruited from the general population through social media advertisements. The study will be carried out for six months, from baseline data collection, follow-up midline data collection, and end-line data collection for outcome measure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intermittent energy restricted (IER) group:
  IER group will receive 5:2 diet pattern (5 day without energy restriction and 2 days with 75% energy restriction, net weekly energy deficit ~25%)
  Interventions: Behavioral: Intermittent energy restriction (IER) : 5:2 diet pattern; Behavioral: Continuous energy restricted (CER) group
- Calorie Restricted Diet (CER) (Active Comparator): Continuous energy restricted (CER) group:
  CER group with a low-calorie diet (daily energy deficit ~25%) over the course of six months.
  Interventions: Behavioral: Intermittent energy restriction (IER) : 5:2 diet pattern; Behavioral: Continuous energy restricted (CER) group

INTERVENTIONS:
Behavioral: Intermittent energy restriction (IER) : 5:2 diet pattern — Participants in the IER group will be provided menus on fasting day that provide ~25% of the individual energy requirement (400 kcal/day for females and 600 kcal/day for males) that means ~75% energy restriction per week (Sundfør et al., 2018; Svendsen, 2018; Templeman, Gonzalez, Thompson, & Betts, 2020). The recommended fasting day may be on two non-consecutive days (Mondays and Thursdays) per week and remaining five days of the week will be based on the usual diet plan. All participants will be instructed to complete all food by 12 pm and then fast until 8 am the following day (Svendsen, 2018).Thus, the weekly average calorie intake will correspond to ~75% of the normal energy requirements. They will receive a diet plan that recommended ~50 gm protein/day from chicken breast, lean meat, lean fish, fat-free yogurt, cottage cheese, egg or legumes, and vegetables to increase satiety on fasting days.
  Other Names: Intermittent fasting
Behavioral: Continuous energy restricted (CER) group — Participants in the CER group will be advised to reduce total energy intake to 1200-1550 kcal in all seven days a week. They will be provided diet plan calculated in relation to each person's estimated energy requirements. Menus will be divided into breakfast, lunch, dinner, and snacks in line with their individualized energy recommendations. They will be requested to consume ~75% of the individual energy requirements daily (25% energy restriction of calculated baseline energy requirements daily) over six months. Thus, the overall energy restriction will similar between the groups at an estimated reduction of 25% of requirements. Participants will be randomized in a 1:1 ratio, and assigned to an intermittent or continuous energy restriction group randomly.
  Other Names: low calorie diet

SUMMARY:
Obesity remains a major public health challenge. Intermittent fasting continues to gain popularity compared to continuous energy restriction as a weight-loss approach for cardiometabolic health. Studies to date comparing intermittent energy restriction (IER) and continuous energy restriction (CER) have not been investigated on weight loss and cardiometabolic risk markers in low-income countries like Nepal. The main objective of this study is to compare the effectiveness of IER versus CER diet on weight loss and cardiometabolic risk markers over the course of six months among overweight/obese Nepalese population.

This study will adopt a parallel arm, open-label, randomized control trial design. The study duration will be six months from baseline to endline. A total of 112 overweight and obese participants, aged 18-64 years, with waist circumference >90 cm (men) and >80 cm (women) will be enrolled in the study. Interested participants will be approached through social media and consecutively enrolled and assigned to either IER group (n=56) or CER group (n=56) randomly. Participants will be provided Mediterranean pattern dietary intervention including two groups: IER group will receive 5:2 diet pattern (5 day without energy restriction and 2 days with 75% energy restriction, net weekly energy deficit ~25%), and CER group with a low-calorie diet (daily energy deficit ~25%) over the course of six months. Both IER and CER group will be provided personalized diet plan, portion size, nutrition counseling focus on dietary guidance, motivational strategies, and personal goal setting for behavior change with educational materials. Baseline data will be collected using a structured questionnaire and the biochemical tests will be done. Baseline data will be collected at the time of enrollment, midline in three months, and end-line data collection in six months. The primary outcome of this study will be the change in weight loss between IER and CER groups. The secondary outcome measure will be to evaluate changes in nutritional composition, eating behavior, and cardiometabolic risk markers between IER and CER group over six months. Data will be entered using Epidata Software and transferred to the Stata/MP version 14.1 for further analysis. Data will be analyzed using an intention-to-treat basis. Independent t-test and, repeated measures ANOVA will be used to estimate changes between-group comparisons. The significance level will be assumed at p<0.05

DETAILED DESCRIPTION:
Overweight and obesity remain a major chronic health problem globally. The development of overweight and obesity is associated with various comorbidities including cardiovascular disease (CVD), dyslipidemia, hypertension, insulin resistance, certain cancers, and sleep apnea. Obesity is a strong modifiable risk factor for CVD, the leading cause of death worldwide. Dietary management is a cornerstone in the prevention, treatment, and control of overweight and obesity, CVD, and metabolic risk factors. Healthy dietary habits reduce the risk of several chronic lifestyle-related diseases as well as meet the demand for essential nutrients to the body to keep healthy.

Many dietary guidelines for the management of overweight and obesity in the general population recommended the reduction of body weight through calorie restriction, increase energy expenditure or followed both approaches. The most common method of weight loss has been daily, or continuous energy restriction (CER), which involves individuals restricting their energy restriction on daily basis by anywhere between 15-60%. Although CER is the most widely recommended calorie restriction approach for body weight loss and prevention of overweight and obesity, recent years have seen a surge in popularity of eating patterns including intermittent energy restriction (IER) as an alternative to CER due to its less restrictive nature and potential for higher rates of adherence. IER is an alternative weight loss method that may prove useful for individuals who find continued energy restriction difficult to maintain. Recent studies have shown IER to be comparable to CER in achieving weight loss in overweight and obese populations with the mean weight loss being 3-5 kg over 20 weeks. IER is considered to be effective for the management of obesity because IER requires the individual to focus on the energy-restricted for defined days during the week which is potentially more feasible than the standard approach of CER which is associated with poor compliance, and IER diet pattern have many beneficial metabolic effects achieved with weight loss and energy restriction when the person is no undergo negative energy balance.

Many peoples are worried about their increased body weight due to obesity-related adverse outcomes including coronary heart disease, type 2 diabetes, and metabolic disorder. There is a knowledge gap of evidence-based dietary patterns used for weight loss diet plan in the Nepalese context. The effectiveness IER using a 2-day severe energy-restricted strategy with 5 days of habitual eating pattern compared to CER has not been yet investigated within the Nepalese population. Therefore, the investigators intended to investigate the effectiveness of an IER diet using 2-day severe energy-restricted with 5 days of habitual eating pattern compared to a CER diet over six months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or above with body mass index (BMI) >25 kg/m2
* Those who give consent to participate in our intervention study

Exclusion Criteria:

* Those who are pregnant women, lactating women, or planning to become pregnant during the course of study.
* Those who are severely ill or more than two comorbidities such as major psychiatric disorders, previous gastric surgery, haematological disorders, insomnia, acute excerabation of chronic obstructive pulmonary disease, asthma, respiratorty tract infections, and diabetes patients if treated with insulin or hypoglycemic agents.
* Those who have any plan to migrate from the study area for at least three months
* Use of anti-obesity drugs or other drugs affecting body weight
* Eating disorder, alcohol or drug abuse that could contribute to difficulties with study procedures

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Body weight | 3 months
  The primary outcome of this study will be the change in reduction of body weight between IER diet using 2-day severe energy-restricted with 5 days of habitual eating pattern compared to a CER diet over three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Dev Ram Sunuwar, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
This is a study protocol, so we don't have any data yet.

REFERENCES:
- [Background] Templeman I, Gonzalez JT, Thompson D, Betts JA. The role of intermittent fasting and meal timing in weight management and metabolic health. Proc Nutr Soc. 2020 Feb;79(1):76-87. doi: 10.1017/S0029665119000636. Epub 2019 Apr 26. PMID 31023390
- [Result] Sundfor TM, Svendsen M, Tonstad S. Effect of intermittent versus continuous energy restriction on weight loss, maintenance and cardiometabolic risk: A randomized 1-year trial. Nutr Metab Cardiovasc Dis. 2018 Jul;28(7):698-706. doi: 10.1016/j.numecd.2018.03.009. Epub 2018 Mar 29. PMID 29778565
- [Result] Pinto AM, Bordoli C, Buckner LP, Kim C, Kaplan PC, Del Arenal IM, Jeffcock EJ, Hall WL. Intermittent energy restriction is comparable to continuous energy restriction for cardiometabolic health in adults with central obesity: A randomized controlled trial; the Met-IER study. Clin Nutr. 2020 Jun;39(6):1753-1763. doi: 10.1016/j.clnu.2019.07.014. Epub 2019 Jul 30. PMID 31409509
- [Result] Sundfor TM, Tonstad S, Svendsen M. Effects of intermittent versus continuous energy restriction for weight loss on diet quality and eating behavior. A randomized trial. Eur J Clin Nutr. 2019 Jul;73(7):1006-1014. doi: 10.1038/s41430-018-0370-0. Epub 2018 Dec 4. PMID 30514879
- [Result] Poirier P, Giles TD, Bray GA, Hong Y, Stern JS, Pi-Sunyer FX, Eckel RH; American Heart Association; Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Obesity and cardiovascular disease: pathophysiology, evaluation, and effect of weight loss: an update of the 1997 American Heart Association Scientific Statement on Obesity and Heart Disease from the Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2006 Feb 14;113(6):898-918. doi: 10.1161/CIRCULATIONAHA.106.171016. Epub 2005 Dec 27. PMID 16380542
- [Result] Rynders CA, Thomas EA, Zaman A, Pan Z, Catenacci VA, Melanson EL. Effectiveness of Intermittent Fasting and Time-Restricted Feeding Compared to Continuous Energy Restriction for Weight Loss. Nutrients. 2019 Oct 14;11(10):2442. doi: 10.3390/nu11102442. PMID 31614992
- [Result] Schubel R, Nattenmuller J, Sookthai D, Nonnenmacher T, Graf ME, Riedl L, Schlett CL, von Stackelberg O, Johnson T, Nabers D, Kirsten R, Kratz M, Kauczor HU, Ulrich CM, Kaaks R, Kuhn T. Effects of intermittent and continuous calorie restriction on body weight and metabolism over 50 wk: a randomized controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):933-945. doi: 10.1093/ajcn/nqy196. PMID 30475957
- [Result] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Result] Seimon RV, Roekenes JA, Zibellini J, Zhu B, Gibson AA, Hills AP, Wood RE, King NA, Byrne NM, Sainsbury A. Do intermittent diets provide physiological benefits over continuous diets for weight loss? A systematic review of clinical trials. Mol Cell Endocrinol. 2015 Dec 15;418 Pt 2:153-72. doi: 10.1016/j.mce.2015.09.014. Epub 2015 Sep 16. PMID 26384657
- [Result] Harvie M, Wright C, Pegington M, McMullan D, Mitchell E, Martin B, Cutler RG, Evans G, Whiteside S, Maudsley S, Camandola S, Wang R, Carlson OD, Egan JM, Mattson MP, Howell A. The effect of intermittent energy and carbohydrate restriction v. daily energy restriction on weight loss and metabolic disease risk markers in overweight women. Br J Nutr. 2013 Oct;110(8):1534-47. doi: 10.1017/S0007114513000792. Epub 2013 Apr 16. PMID 23591120
- [Result] Antoni R, Johnston KL, Collins AL, Robertson MD. Intermittent v. continuous energy restriction: differential effects on postprandial glucose and lipid metabolism following matched weight loss in overweight/obese participants. Br J Nutr. 2018 Mar;119(5):507-516. doi: 10.1017/S0007114517003890. PMID 29508693
- [Result] Carter S, Clifton PM, Keogh JB. The effects of intermittent compared to continuous energy restriction on glycaemic control in type 2 diabetes; a pragmatic pilot trial. Diabetes Res Clin Pract. 2016 Dec;122:106-112. doi: 10.1016/j.diabres.2016.10.010. Epub 2016 Oct 19. PMID 27833048
- [Result] Harvie M, Howell A. Potential Benefits and Harms of Intermittent Energy Restriction and Intermittent Fasting Amongst Obese, Overweight and Normal Weight Subjects-A Narrative Review of Human and Animal Evidence. Behav Sci (Basel). 2017 Jan 19;7(1):4. doi: 10.3390/bs7010004. PMID 28106818